CLINICAL TRIAL: NCT05177224
Title: In Vivo Study of the Dual Mobility Cup Stability and Mobility Using Ultrasound Imaging
Brief Title: Ultrasound Imaging of Dual Mobility Cup
Acronym: USDMC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL21_0884
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Dual Mobility Cups
Keywords: dual mobility cup; liner; motion analysis; ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with dual mobility cup (Experimental)
  Interventions: Other: Ultrasound acquisitions to define liner position during movements

INTERVENTIONS:
Other: Ultrasound acquisitions to define liner position during movements — Ultrasound acquisition of the dual mobility cup will be performed before and after movement. Acquisitions will be performed on the groin area.
  Movement will be performed 3 times and are:
  * Walking
  * Knee-bending
  * Standing up
  * Stair climbing Movement acquisition of the lower limb will be performed using reflective markers placed on the skin. The movements will be recorded using motion capture system (infrared cameras). The load applied by the patients on the ground when doing these movements will be recorded with a force plate.

SUMMARY:
The concept of dual mobility cup (DMC), developed in the 1970s by Gilles Bousquet, allows a greater motion and a better stability of the implants, reducing the prosthetic dislocations frequency in at-risk populations. This type of prosthesis has a small-diameter head that ensures a low wear rate and a large-diameter head, with a polyethylene liner, to increase prosthetic stability. This prosthesis has survival rates comparable to those found with conventional prostheses. However, actually, its in vivo behaviour has not yet been established, leading orthopaedic surgeons to keep this concept for patients with a high risk of dislocation (elderly subjects, neurological pathologies, spinal pathologies, falls, etc.). To date, no in vivo studies have been carried out - non-invasively and dynamically - to understand the biomechanical behaviour and the stability properties of the dual mobility cup implanted in patients.

The objective of this study is to visualize and quantify the in vivo movement of the polyethylene liner using 3D ultrasound imaging. The second objective is to obtain in vivo data (using the motion analysis system and the force platform) allowing the use of a musculoskeletal model to improve the understanding of the prosthetic dislocation phenomenon.

Participants will carry out daily life activities (walk, chair up, etc.). During this study, liner ultrasound acquisitions and motion analysis of the lower limb will be performed, thanks to a movement analysis system composed of cameras coupled to a force platform.

Hip kinematics will be obtained from the motion analysis data and will be based on the model of Leardini et al. 2007. The position of the liner and liner plane will be determined using 3D ultrasound data. The abduction and anteversion motion of the liner plane will be measured relative to the pelvic landmark.

ELIGIBILITY:
Inclusion Criteria:

* Patient having signed a free and informed consent
* Being affiliated or benefiting from a social security system
* Having dual mobility cup for at least 1 year
* Outside of a period of exclusion from the national file of persons undergoing biomedical research
* Age greater than or equal to 50 years
* Of a cognitive level compatible with oral communication, the respect of instructions and the understanding of the gestures carried out

Exclusion Criteria:

* Persons who are not physically able to perform tests
* Persons currently participating in another research project with an exclusion period
* Persons of full age under legal protection or unable to express their consent
* Pregnant or breast-feeding women (Article L1121-5 of the Public Health Code (CSP))
* Persons deprived of their liberty by a judicial or administrative decision, persons under psychiatric care and persons admitted to a health or social institution for purposes other than research

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Liner position using ultrasound | At inclusion (At least one year after surgery)
  The liner position and liner plane are defined using 3D ultrasound data. Abduction and anteversion motion of the liner plane are measured relative to the pelvic landmark.

SECONDARY OUTCOMES:
Hip kinematics using motion analysis | At inclusion (At least one year after surgery)
  Hip kinematics is obtained using motion analysis data and based on the Leardini et al. model (Leardini et al. 2007). The pelvic benchmark will be determined according to the ISB recommendations (Derrick et al. 2020).
Forces and moments during movements | At inclusion (At least one year after surgery)
  Forces and moments during movement are measured using a force plate.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hôpital Lyon Sud - Service de Chirurgie Orthopédique, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided